CLINICAL TRIAL: NCT05474300
Title: Retrospective Evaluation of the Effect of Slope Time in PCV Mode on Mechanical Power Calculation and Oxygenation in Covid-19 ARDS Patients.
Brief Title: Effect of Slope Time in PCV Mode on Mechanical Power Calculation and Oxygenation in Covid-19 ARDS Patients.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Bakirkoy Dr. Sadi Konuk Research and Training Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2022/209
Record Dates: First submitted 2022-07-25; First posted 2022-07-26 (Actual); Last update posted 2022-08-03 (Actual); Status verified 2022-08

CONDITIONS: COVID-19 Pneumonia; COVID-19 Acute Respiratory Distress Syndrome
Keywords: Tslope; Pressure controlled ventilation; mechanical ventilation
MeSH Terms: interventions — Respiration, Artificial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Covid-19 ARDS patients on PCV mode: No Intervention
  Interventions: Other: mechanical ventilation

INTERVENTIONS:
Other: mechanical ventilation — Pressure controlled ventilation mode on mechanical ventilation

SUMMARY:
The investigators are planning to investigate the effect of each 5% slope time change on mechanical power and SPO2 of the patients with Covid 19 ARDS diagnosis which are on mechanical ventilation PCV mode support.

DETAILED DESCRIPTION:
In this study, with inspiration/expiration 1:2 and 1:1 time ratios in pressure controlled ventilation mode with different slope times mechanical power will be calculated in covid ARDS patients. In this way, the effect of every 5% slope time change in PCV on mechanical power and SPO2 will be investigated.

ELIGIBILITY:
Inclusion Criteria:

* adult patients with Covid-19 Acute Respiratory Distress Syndrome (ARDS) diagnosis
* intubated Covid-19 ARDS patients
* Covid-19 ARDS patients on mechanical ventilator support

Exclusion Criteria:

* heart failure disease
* Chronic Obstructive Pulmonary Disease (COPD)
* hemodynamically unstable patients
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with Covid-19 ARDS diagnosis which has been admitted to intensive care unit, intubated and are on PCV mode on mechanical ventilation support will be included in the study.
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2022-06-06 (Actual); Primary Completion 2022-08-06 (Estimated); Study Completion 2022-08-30 (Estimated)

PRIMARY OUTCOMES:
mechanical power | 100 minutes
  Mechanical power calculated by Becher et al. comprehensive formula (MPpcv(slope)) and Trinkle, Christine A et al lineer model mechanical power formula (MPLM).

CONTACTS AND LOCATIONS:
Overall Officials: sinan asar, M.D, Study Director — intensive care supspecialist
Locations (1):
- Bakırköy Dr sadi konuk Education hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Becher T, van der Staay M. Calculation of mechanical power for pressure-controlled ventilation: author's reply. Intensive Care Med. 2019 Oct;45(10):1498-1499. doi: 10.1007/s00134-019-05742-7. Epub 2019 Aug 20. No abstract available. PMID 31432217
- [Result] Trinkle CA, Broaddus RN, Sturgill JL, Waters CM, Morris PE. Simple, accurate calculation of mechanical power in pressure controlled ventilation (PCV). Intensive Care Med Exp. 2022 May 30;10(1):22. doi: 10.1186/s40635-022-00448-5. PMID 35644896